CLINICAL TRIAL: NCT02184832
Title: Dietary Intake of Tryptophan and Metformin Response
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Geoffrey Walford, MD, Instructor in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P001226
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Metformin Response; Fasting Glucose; Tryptophan Concentration; Metformin Concentration; Diet Tolerability
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low tryptophan diet (Experimental): 2 days of a low tryptophan diet
  Interventions: Drug: Metformin; Other: Low tryptophan diet
- High tryptophan diet (Experimental): 2 days of a high tryptophan diet
  Interventions: Drug: Metformin; Other: High tryptophan diet

INTERVENTIONS:
Drug: Metformin — 2 doses of 500 mg metformin given approximately 12 hrs apart
Other: Low tryptophan diet
  Arms: Low tryptophan diet
Other: High tryptophan diet
  Arms: High tryptophan diet

SUMMARY:
This study will examine the influence of dietary intake of tryptophan on response to metformin. The investigators hypothesize that dietary tryptophan alteration will influence metformin response.

ELIGIBILITY:
Inclusion Criteria:

1. healthy adult male or non-pregnant female volunteers (age 20-40)
2. able and willing to give consent

Exclusion Criteria:

1. Age less than 20 or greater than 40
2. Women who are pregnant, nursing, or at risk of becoming pregnant
3. Body mass index (BMI) less than 20 or greater than 28
4. Changes of more than 5 pounds in weight (increase or decrease) during the month prior to enrollment in the study
5. Participation in more than 300 minutes of exercise per week during the month prior to enrollment in the study
6. Known diabetes or pre-diabetes (based on prior diagnoses, use of medications to lower glucose; or fasting blood glucose > 100mg/dL at screening)
7. Untreated hypertension (defined as systolic blood pressure > 140mmHg and diastolic blood pressure > 90mmHg)
8. Current or past mood disorder, including major depression, anxiety, or bipolar disorder
9. Conditions causing intestinal malabsorption, including celiac disease or a history of intestinal or gastric bypass surgery
10. History of liver disease and/or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 3 times upper limit of normal (ULN)
11. Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation
12. Currently taking or intending to take during the study duration any medication known to affect glycemic parameters, such as glucocorticoids, growth hormone, or fluoroquinolones
13. Use of medications and herbal or vitamin supplements during the study
14. Contraindications to safe use of metformin, including planned radiologic or angiographic study requiring contrast within one week of the study completion
15. Objection to taking metformin
16. Participation in any other interventional study during the study duration
17. Use of nicotine-containing products, including inhaled, chewed, or patches during the study.
18. Use of drugs of abuse.
19. Restrictions that prevent adherence to standardized meals or unwillingness to adhere to a pre-specified meal plan, including abstinence from alcohol and limitation of caffeine intake to one drink daily.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
change in fasting glucose | 2 days

SECONDARY OUTCOMES:
change in tryptophan concentration | 2 days

OTHER OUTCOMES:
tolerability of dietary tryptophan alteration | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Walford, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States